CLINICAL TRIAL: NCT00458549
Title: Prostate Cancer Prevention by n-3 Unsaturated Fatty Acids
Brief Title: Polyunsaturated Fatty Acids in Treating Patients With Prostate Cancer Undergoing Prostate Biopsy and/or Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jose A. Halperin, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 03-116; R01CA101034 (NIH); P30CA006516 (NIH)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fatty Acids, Omega-3; Biopsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omega-3 fatty acids (Experimental): omega-3 fatty acids Oral 8g once a day for 21 days prior to (biopsy) surgery
  Interventions: Dietary Supplement: omega-3 fatty acids; Procedure: biopsy
- Corn Oil (Placebo Comparator): Oral 8g once a day for 21 days prior to (biopsy) surgery
  Interventions: Procedure: biopsy

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acids — omega-3 fatty acids Oral 8g once a day for 21 days prior to (biopsy) surgery
  Other Names: OmegaRx
  Arms: omega-3 fatty acids
Procedure: biopsy

SUMMARY:
RATIONALE: Polyunsaturated fatty acids are important for normal growth and development. One type, called omega-3 fatty acids (found in fish, fish oil, and some other foods), may affect the growth of prostate cancer.

PURPOSE: This randomized clinical trial is studying polyunsaturated fatty acids in treating patients with prostate cancer undergoing prostate biopsy and/or surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare fatty acid analysis of red blood cells, levels of eIF2α phosphorylation, and tumor differentiation grade, as measured by Gleason score, in patients undergoing prostate biopsy. (Part 1)
* Determine if neoadjuvant n-3 polyunsaturated fatty acids (PUFAs) induce phosphorylation of eIF2α in these patients. (Part 2)
* Compare eIF2α phosphorylation, Gleason score, and the time to prostate-specific antigen failure in prostate tumor samples obtained from the Gelb Center of the Dana-Farber Cancer Institute prostate tissue repository. (Part 3)

OUTLINE: This is a prospective study, followed by a randomized, double-blind, placebo-controlled study, followed by a retrospective study.

* Part 1: Patients undergo tumor biopsy and blood sample collection at baseline. Samples are analyzed by gas-liquid chromatography for determination of n-3 and n-6 polyunsaturated fatty acid (PUFA) red cell membrane concentrations. Biopsy samples are analyzed for eIF2α phosphorylation by immunohistochemistry. Some patients proceed to part 2.
* Part 2: Patients undergo blood sampling as in part 1 with additional tumor and blood collection on day 28. Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral n-3 PUFAs (fish oil) once daily for 28 days prior to tumor resection.
  * Arm II (control): Patients receive oral n-6 PUFAs (corn oil) once daily for 28 days prior to tumor resection.
* Part 3: Tumor samples and associated pathology data (Gleason score) and clinical data (PSA values and patient's outcome) are obtained from a prostate tissue repository at the Gelb Center of the Dana-Farber Cancer Institute. Samples are analyzed to correlate eIF2α phosphorylation, Gleason scores, and time to PSA failure.

PROJECTED ACCRUAL: A total of 600 patients and 1,000 stored tissue samples will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing an outpatient prostate biopsy independently indicated by a physician.
* Patients will be selected from the population initially studied with a prostate biopsy for possible prostate cancer

  * sub-group without evidence of cancer
  * sub-group with advanced prostate cancer beyond the currently accepted criteria for surgical treatment,
  * sub-group with indication of radical prostatectomy
* Patients will be recruited from the population of patients from Brigham and Women's Hospital for surgery referred from other institutions/doctors where their biopsy was taken and the diagnosis of prostate cancer was originally made. These patients are not eligible for Aim 1 but will enter the randomized trial (Aim 2 with baseline)

Exclusion Criteria:

* Prostate biopsy patients who do not accept and sign an informed consent form to

  * donate ten ml of blood for fatty acid analysis in red blood cells
  * allow their prostate biopsy to be analyzed as discarded pathological material
  * authorize access to their hospital clinical information for follow up studies
* Patients with a current diagnosis of a condition that might interfere with the measurements of fatty acids in red blood cell membranes such as severe anemia (less than 9g/100m1% hemoglobin

  -- Or
* Diseases of lipid metabolism such as familial dyslipoproteinemia, liver cirrhosis, advanced renal failure, and malabsorption syndrome.
* Exclude from this study patients from (indication of radical prostatectomy) who refuse the surgical recommendation or schedule surgery at a location other than Brigham and Women's Hospital.
* Patients who are not able to complete the full program will not be taken into consideration in the final data analysis.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2003-05-27 (Actual); Primary Completion 2009-05-14 (Actual); Study Completion 2012-05-01 (Actual)

PRIMARY OUTCOMES:
Level of eIF2α phosphorylation and Gleason score in prostate biopsy samples (Part 1) | 21 Days
Change in phosphorylation level of eIF2α before and after n-3 polyunsaturated fatty acid supplementation (Part 2) | 21 Days

SECONDARY OUTCOMES:
Relapse-free survival (Part 2) | Time between surgery and the time of PSA failure 6 months and 9 months
  detectable (> 0.1ng/m1) values following an undetectable level

CONTACTS AND LOCATIONS:
Overall Officials: Jose A. Halperin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No